CLINICAL TRIAL: NCT02394873
Title: A Phase 1 Clinical Study to Evaluate the Safety of Allogeneic Adipose-derived Stem Cells in the Subjects With Deep Second-degree Burn Wound
Brief Title: A Study to Evaluate the Safety of ALLO-ASC-DFU in the Subjects With Deep Second-degree Burn Wound
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-BI-101
Record Dates: First submitted 2015-03-06; First posted 2015-03-20 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Burn
Keywords: Deep Second-Degree Burn Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALLO-ASC-DFU (Experimental)
  Interventions: Biological: ALLO-ASC-DFU

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Dressing for second-degree burn wound.

SUMMARY:
This is a phase I study to evaluate the safety of ALLO-ASC-DFU for the treatment of deep second-degree burn wound patients. ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a burn.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age and older.
2. Subjects who have deep second-degree burn ≥100 cm^2.
3. Negative for urine beta-HCG for women of childbearing age.
4. Subject is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who have been enrolled in another clinical study within 30 days of screening.
2. Subjects who are allergic or have a hypersensitive reaction to bovine-derived proteins or fibrin glue.
3. Subjects who are receiving steroids, immunosuppressive, or anticoagulant.
4. Subjects with active infection.
5. Subjects with hemorrhagic and hemocoagulative disease
6. Subjects who are unwilling to use an "effective" method of contraception during the study.
7. Subjects who have a history of malignant tumor within the last five years, or is currently undergoing.
8. Subjects who are pregnant or breast-feeding.
9. Subjects who are considered to have a significant disease which can impact the study by the investigator
10. Burn wound is present on any part of the face.
11. Subjects who have a history of surgery for malignant tumor within the last five years (except carcinoma site).
12. Subjects who are considered not suitable for the study by the investigator.
13. Subjects who are not able to understand the objective of this study or to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 4 weeks

SECONDARY OUTCOMES:
Time to reach re-epithelialization of wound | 1, 2, 4 weeks
  Evaluation of the improvement of wound measured by time to reach re-epithelialization of wound
Vancouver Burn Scar Scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wook Chun, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym university Medical Center, Seoul, South Korea